CLINICAL TRIAL: NCT00374803
Title: A 12-month, Prospective, Randomized, Single Center, Open Label Pilot Study to Evaluate the Safety and Efficacy of Myfortic in Combination With Tacrolimus and Thymoglobulin in Early Corticosteroid Withdrawal
Brief Title: Study of Myfortic in Combination With Tacrolimus and Thymoglobulin in Early Corticosteroid Withdrawal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Rita Alloway, PharmD, FCCP, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyforticINVINT
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Kidney; Transplant; Corticosteroid; Myfortic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolic Acid (Myfortic) Preload (Experimental): Mycophenolic Acid (Myfortic) 1080 mg twice daily (2160 mg/day) for two weeks, followed by 720 mg twice daily (1440 mg/day) thereafter
  Interventions: Drug: Mycophenolic Acid (Myfortic)
- Mycophenolic Acid (Myfortic) Standard (Active Comparator): Mycophenolic Acid (Myfortic) 720 mg twice daily (1440 mg/day).
  Interventions: Drug: Mycophenolic Acid (Myfortic)

INTERVENTIONS:
Drug: Mycophenolic Acid (Myfortic) — * Group 1: Mycophenolic Acid (Myfortic) 1080 mg twice daily (2160 mg/day) for two weeks, followed by 720 mg twice daily (1440 mg/day) thereafter
  * Group 2: Mycophenolic Acid (Myfortic) 720 mg twice daily (1440 mg/day).
  Other Names: mycophenolic acid enteric coated

SUMMARY:
To determine the safety and efficacy of a new formulation of Myfortic in combination with tacrolimus and thymoglobulin.

DETAILED DESCRIPTION:
Evaluate the safety and efficacy of Myfortic in combination with tacrolimus and anti-thymocyte globulin in an early corticosteroid withdrawal protocol. Secondary objective is to determine the pharmacokinetic-pharmacodynamic profile of Myfortic in a corticosteroid withdrawal protocol.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 75 years of age.
* Patients who are primary or repeat cadaveric, living unrelated or non-HLA identical living related donor renal transplant recipients.

Exclusion Criteria:

* Patient previously received or is receiving an organ transplant other than kidney.
* Primary or re-transplant from human leukocyte antigen (HLA)-identical living donor.
* Recipient or donor is known to be seropositive for hepatitis C virus (HCV), hepatitis B virus (HBV), or human immunodeficiency virus (HIV).
* Uncontrolled concomitant infection or other unstable medical condition.
* Patients that received an investigational drug in the 30 days prior to transplant.
* Known hypersensitivity to tacrolimus, mycophenolate mofetil (MMF), enteric-coated mycophenolic acid, rabbit anti-thymocyte globulin, or corticosteroids.
* Receiving chronic steroid therapy at the time of transplant.
* History of malignancy in last 5 years.
* Pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Alloway, PharmD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center, 45 patients consecutively enrolled. Patients were randomized into two groups: (group 1) will be receive 2160 mg/day for two weeks, followed by 1440 mg/day thereafter, and (group 2) will receive 1440 mg/day for the duration of the study.
Groups:
- Myfortic 1080mg BID, 720mg BID: Myfortic 1080 mg twice daily (2160 mg/day) for two weeks, followed by 720 mg twice daily (1440 mg/day) thereafter
- Myfortic 720 mg Twice Daily: Myfortic 720 mg twice daily (1440 mg/day).
Period: Overall Study
Arm/Group | Myfortic 1080mg BID, 720mg BID | Myfortic 720 mg Twice Daily
Started | 22 | 23
Completed | 22 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myfortic 1080mg BID, 720mg BID | Myfortic 720 mg Twice Daily | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 55 (13) | 52 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All Biopsy Proven Acute Rejection.
Description: Treatment efficacy, defined as the incidence of all biopsy proven acute rejection. Biopsy was proven with tissue samples collected on patients with elevated serum creatinine
Time Frame: 12 months
Measure: Number; unit: Participants
Groups:
- Mycophenolic Acid Loading Group: Thymoglobulin 1.5 mg/kg/dose x 4 doses on days 0, 2, 4 and 6, Tacrolimus 0.1 mg/kg/day divided twice daily, 7 days corticosteroid taper, and Myfortic 1080 mg twice daily (2160 mg/day) for two weeks, followed by 720 mg twice daily (1440 mg/day) thereafter
- Mycophenolic Acid No Load Group: Thymoglobulin 1.5 mg/kg/dose x 4 doses on days 0, 2, 4 and 6, Tacrolimus 0.1 mg/kg/day divided twice daily, 7 days corticosteroid taper, and Myfortic 720 mg twice daily (1440 mg/day)
Arm/Group | Mycophenolic Acid Loading Group | Mycophenolic Acid No Load Group
Number analyzed (Participants) | 22 | 23
Participants | 1 | 4

2. Secondary Outcome: Patient and Allograft Survival 12 Months
Description: Patient and allograft survival at 12 months post-transplant. Allograft survival is different from rejection. An allograft can have rejection, but the allograft can still have survival. If an allograft fails and is no longer functioning this would be considered allograft failure and non-survival.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Mycophenolic Acid (Myfortic) Preload: Mycophenolic Acid (Myfortic) 1080 mg twice daily (2160 mg/day) for two weeks, followed by 720 mg twice daily (1440 mg/day) thereafter
  Mycophenolic Acid (Myfortic): • Group 1: Mycophenolic Acid (Myfortic) 1080 mg twice daily (2160 mg/day) for two weeks, followed by 720 mg twice daily (1440 mg/day) thereafter
  • Group 2: Mycophenolic Acid (Myfortic) 720 mg twice daily (1440 mg/day).
- Mycophenolic Acid (Myfortic) Standard: Mycophenolic Acid (Myfortic) 720 mg twice daily (1440 mg/day).
  Mycophenolic Acid (Myfortic): • Group 1: Mycophenolic Acid (Myfortic) 1080 mg twice daily (2160 mg/day) for two weeks, followed by 720 mg twice daily (1440 mg/day) thereafter
  • Group 2: Mycophenolic Acid (Myfortic) 720 mg twice daily (1440 mg/day).
Arm/Group | Mycophenolic Acid (Myfortic) Preload | Mycophenolic Acid (Myfortic) Standard
Number analyzed (Participants) | 22 | 23
participants
  Patient Survival | 22 | 23
  Allograft Survival | 22 | 22

3. Secondary Outcome: Renal Function at 12 Months
Description: Renal function measured by serum creatinine (SCr) at 12 months post-transplant
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mycophenolic Acid Loading Group | Mycophenolic Acid No Load Group
Number analyzed (Participants) | 22 | 22
mg/dL | 1.36 (0.4) | 1.5 (1.0)

4. Secondary Outcome: Incidence of Post Transplant Infections
Description: Incidence of post transplant infections that resulted in hospitalization
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Mycophenolic Acid Loading Group | Mycophenolic Acid No Load Group
Number analyzed (Participants) | 22 | 23
participants | 4 | 4

5. Secondary Outcome: GI Toxicities
Description: Hospitalizations due to Gastrointestinal (GI) toxicities of mycophenolic acid enteric coated (Myfortic)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Mycophenolic Acid Loading Group | Mycophenolic Acid No Load Group
Number analyzed (Participants) | 22 | 23
participants | 5 | 4

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Mycophenolic Acid Loading Group | Mycophenolic Acid No Load Group
Serious Adverse Events (participants affected / at risk) | 4/22 | 14/23
Other Adverse Events (participants affected / at risk) | 17/22 | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolic Acid Loading Group (N=22) | Mycophenolic Acid No Load Group (N=23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (4) | 4 (4)
Fever (General disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Creatinine Increased (Investigations) | 0 (0) | 4 (8)
Acute Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Kidney Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Worsening Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehiscence with evisceration (Surgical and medical procedures) | 0 (0) | 1 (2)
Coronary Artery Bypass (Cardiac disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Altered Mental Status (Nervous system disorders) | 0 (0) | 1 (1)
Post-transplant lymphoproliferative disorder (PTLD) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Mycophenolic Acid Loading Group (N=22) | Mycophenolic Acid No Load Group (N=23)
Diarrhea (Gastrointestinal disorders) | 4 | 4
Wound dehiscence (Skin and subcutaneous tissue disorders) | 2 | 0
CMV Viremia (Immune system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 9 | 10/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No